CLINICAL TRIAL: NCT00028509
Title: Assessment of Clinical and Neuroradiologic Evidence of Methotrexate Leukoencephalopathy in Children Treated on POG 9605 and 9201
Brief Title: Brain Function in Children Previously Treated on Clinical Trials POG-9605 and POG-9201
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: ACCL0131; COG-ACCL0131 (Other: Children's Oncology Group); NCI-P01-0198; CDR0000069100 (Other: Clinical Trials.gov)
Record Dates: First submitted 2002-01-04; First posted 2003-01-27 (Estimated); Last update posted 2014-02-13 (Estimated); Status verified 2014-02

CONDITIONS: Long-term Effects Secondary to Cancer Therapy in Children; Neurotoxicity
Keywords: neurotoxicity; long-term effects secondary to cancer therapy in children
MeSH Terms: conditions — Neurotoxicity Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: management of therapy complications

SUMMARY:
RATIONALE: Assessing the effects of methotrexate on brain function in children may improve the ability to plan treatment and decrease side effects.

PURPOSE: Clinical trial to compare brain function of children who have been previously treated with methotrexate.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the incidence of neuropsychological abnormalities and leukoencephalopathy in children previously treated with methotrexate on protocols POG-9605 versus POG-9201.

OUTLINE: This is a multicenter study.

More than 3 years after completion of therapy, patients undergo 9 different tests to assess intelligence, memory, learning, attention, concentration, processing of information, functioning, and visual-motor integration. Patients also undergo MRI of the head.

PROJECTED ACCRUAL: A total of 30-54 patients previously treated on protocol POG-9201 will be accrued for this study. A total of 60-108 patients previously treated on protocol POG-9605 will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Previously enrolled on POG-9201 or POG-9605

  * Good prognosis by NCI risk (9201 and 9605 stratum 1)
* Eligible for the therapeutic study
* Completed therapy by 12/31/2000
* No CNS3 at diagnosis
* No relapsed disease

PATIENT CHARACTERISTICS:

Age:

* 1 to 9 at diagnosis

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

Other:

* No Down syndrome

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* See Disease Characteristics

Ages: 1 Year to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Previously enrolled on POG-9201 or POG-9605
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2002-07; Primary Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with severe intelligence deficit as evidenced by either a verbal or performance IQ below 85 | Length of study

SECONDARY OUTCOMES:
Compare the groups for descriptive purposes | Length of study
  Quantitative scales: IQ (WISC III or WPPSI-R, depending on the age of the child), Wide Range Assessment of Memory and Learning (4 subscales), Conner's Continuous Performance Test (Attention/Concentration), Woodcock Johnson Revised Processing Speed Cluster, NEPSP Tower Tests (Executive Functioning), and VSI (Visual-Motor Integration).

CONTACTS AND LOCATIONS:
Overall Officials: Patricia K. Duffner, MD, Study Chair — Women & Children's Hospital of Buffalo
Locations (26):
- United States (25):
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Stanford Comprehensive Cancer Center - Stanford, Stanford, California
  - University of Miami Sylvester Comprehensive Cancer Center - Miami, Miami, Florida
  - Miami Children's Hospital, Miami, Florida
  - St. Joseph's Cancer Institute at St. Joseph's Hospital, Tampa, Florida
  - Kaplan Cancer Center at St. Mary's Medical Center, West Palm Beach, Florida
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - Rush University Medical Center, Chicago, Illinois
  - CancerCare of Maine at Eastern Maine Medial Center, Bangor, Maine
  - Floating Hospital for Children at Tufts - New England Medical Center, Boston, Massachusetts
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - University of Mississippi Cancer Clinic, Jackson, Mississippi
  - Siteman Cancer Center at Barnes-Jewish Hospital, St Louis, Missouri
  - Hackensack University Medical Center Cancer Center, Hackensack, New Jersey
  - University of New Mexico Cancer Research and Treatment Center, Albuquerque, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - Blumenthal Cancer Center at Carolinas Medical Center, Charlotte, North Carolina
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Oklahoma University Cancer Institute, Oklahoma City, Oklahoma
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - Baylor University Medical Center - Houston, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Midwest Children's Cancer Center, Milwaukee, Wisconsin
- Montreal Children's Hospital at McGill University Health Center, Montreal, Quebec, Canada